CLINICAL TRIAL: NCT02010385
Title: Investigation of the Effects of Obesity Surgery on Appetitive Behaviour - Impact of Gut Hormones
Brief Title: Investigation of the Effects of Obesity Surgery on Appetitive Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Carel le Roux, Prof, PhD, MSc, MRCPath, MRCP, MBChB, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: Le Roux 12 June 12
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Roux-en-Y Bariatric Surgery
Keywords: RYGB; Bariatric surgery; Taste; Reward; Food behaviour; Gut hormones
MeSH Terms: interventions — Octreotide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Octreotide (Active Comparator): One subcutaneous injection - 1 mL
  Interventions: Drug: Octreotide
- Saline (Placebo Comparator): One subcutaneous injection - 1 mL
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Octreotide
  Other Names: Octreotide 100 micrograms/1ml - solution for injection - Hospira - Q64021
  Arms: Octreotide
Drug: Saline
  Other Names: Sodium chloride 0.9% W/V injection BP - Fannin - PL 24598/0002
  Arms: Saline

SUMMARY:
Among all the existing ways to treat obesity (lifestyle, pharmacological), Roux-en-Y gastric bypass (RYGB) surgery is currently the most effective. It results in long term weight loss maintenance, significant remission of obesity-related comorbidities and decreased overall mortality. It also induces changes in gastrointestinal hormones responses, with an increase of anorexigenic hormones GLP-1, and PYY.

Although successful, the mechanisms for RYGB-induced weight loss are not completely understood. The RYGB does result in increased satiation, decreased calorie intake and decreased preferences for sweet and fatty foods. Previous work from our lab has shown using progressive ratio task (PRT) that RYGB specifically decreases the appetitive behaviour for sweet and fat stimuli but not for vegetables. The reasons for this change in appetitive behaviour after the surgery remain unknown. They may be triggered by changes in gut hormones, conditioned taste aversion (negative post-ingestive effects) or changes in serum bile acids levels.

This study aims to assess whether RGYB-induced gut hormone changes contribute to the decrease in appetitive behaviour for sweet and fatty foods observed after the surgery.

This is a double blind controlled study comparing the effect of blocking gut hormones with somatostatin analogue (octreotide) on the appetitive behaviour for sweet-fat candies will be carried out. Appetitive behaviour will be measured using the progressive ratio task.

The investigators hypothesize that blocking the gut hormones in obese patients with RYGB will increase their appetitive behaviour for sweet-fat candies.

ELIGIBILITY:
Inclusion Criteria:

* Gastric bypass surgery since at least 6 months

Exclusion Criteria:

* serious illness
* pregnancy or breast feeding
* more than three alcoholic drinks per day
* substance abuse
* psychiatric illness
* significant longstanding heart disease or heart intervention (for example, patients who have had heart attacks, have pacemakers or have had heart surgery)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Progressive ratio breakpoint | One hour
  In the Progressive ratio task, the participants click a computer mouse in order to obtain a sweet/fat food reward. The effort required to obtain a reward is progressively increased. The breakpoint refers to the point at which the reward value of the food stimulus is lower than the effort necessary to obtain it and the participant stops pressing the button.

SECONDARY OUTCOMES:
Subjective ratings | One hour
  Hunger, fullness, desire in eating and nausea state will be assessed using Visual Analogue Scales (VAS).
Gut hormones level | One hour
  GLP-1, ghrelin, leptin and insulin levels will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Carel le Roux, Pr, MD, Principal Investigator — UCD Conway institute
Locations (1):
- University College Dublin Clinical Research Centre, Dublin, Ireland

REFERENCES:
- [Background] Miras AD, Jackson RN, Jackson SN, Goldstone AP, Olbers T, Hackenberg T, Spector AC, le Roux CW. Gastric bypass surgery for obesity decreases the reward value of a sweet-fat stimulus as assessed in a progressive ratio task. Am J Clin Nutr. 2012 Sep;96(3):467-73. doi: 10.3945/ajcn.112.036921. Epub 2012 Jul 25. PMID 22836034